CLINICAL TRIAL: NCT01041586
Title: US Pilot Safety and Feasibility Study of Bronchoscopic Thermal Vapor Ablation (BTVA) for Lung Volume Reduction in Patients With Heterogeneous Emphysema With Upper Lobe Predominance
Brief Title: Bronchoscopic Thermal Vapor Ablation (BTVA) for Lung Volume Reduction
Acronym: BTVA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uptake Medical Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAPOR-US
Record Dates: First submitted 2009-12-22; First posted 2009-12-31 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: Emphysema; COPD; Lung Volume Reduction; BTVA
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BTVA (Experimental)
  Interventions: Device: BTVA System

INTERVENTIONS:
Device: BTVA System — Unilateral Bronchoscopic Thermal Vapor Ablation for Lung Volume Reduction

SUMMARY:
To assess the safety and efficacy of BTVA for the treatment of patients with heterogeneous upper lobe emphysema.

DETAILED DESCRIPTION:
All subjects meeting the eligibility criteria and who provide written informed consent will be enrolled. Immediately prior to BTVA treatment, an initial bronchoscopy will be performed to evaluate the baseline condition of the airways and to confirm anatomy of the lung segments targeted for BTVA treatment. Up to 3 segments in either the right or left upper lobe will be treated with a vapor dose of 10 calories per gram of lung tissue (10 cal/g). Targeted lobe for treatment will be based on lobar disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 40 and ≤ 75 years old
2. Diagnosis of heterogeneous emphysema with upper lobe predominance
3. FEV1 < 45% predicted
4. TLC > 100% predicted
5. RV > 150% predicted
6. 6-minute walk test > 140 meters
7. mMRC ≥ 2 (mMRC)
8. Non-smoking for 3 months
9. Optimized medical management and completed pulmonary rehabilitation

Exclusion Criteria:

1. Known α-1-antitrypsin deficiency
2. BMI < 15 kg/m2 or > 35 kg / m2
3. History of pneumothorax within previous 18 months
4. History of heart and / or lung transplant, lung volume reduction surgery (LVRS), median sternotomy, bullectomy, and/or lobectomy
5. Respiratory infections or recurring COPD exacerbations > 3 hospitalizations in past 12 months or active infection
6. History of the (EF) ≤ 40%; Stroke; Unstable Myocardial Ischemia; FEV1 < 15% predicted; DLCO < 20% predicted; of pulmonary hypertension; indwelling pacemaker or implantable cardiac defibrillator (ICD); pregnancy or breastfeeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events (serious and non-serious) secondary to the BTVA treatment procedure from initiation of treatment through completion of the six-month follow-up period | 6 months

SECONDARY OUTCOMES:
Radiographic evidence of lung volume reduction (assessed by study site radiologist) and CT scan (assessed by blinded radiologist at CT core lab) | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - John C. Lincoln Hospital, Phoenix, Arizona
  - University of Iowa, Iowa City, Iowa
  - Boston, Massachusetts
  - Swedish Hospital, Seattle, Washington

REFERENCES:
- [Derived] Herth FJ, Ernst A, Baker KM, Egan JJ, Gotfried MH, Hopkins P, Stanzel F, Valipour A, Wagner M, Witt C, Kesten S, Snell G. Characterization of outcomes 1 year after endoscopic thermal vapor ablation for patients with heterogeneous emphysema. Int J Chron Obstruct Pulmon Dis. 2012;7:397-405. doi: 10.2147/COPD.S31082. Epub 2012 Jul 18. PMID 22927751
- [Derived] Snell G, Herth FJ, Hopkins P, Baker KM, Witt C, Gotfried MH, Valipour A, Wagner M, Stanzel F, Egan JJ, Kesten S, Ernst A. Bronchoscopic thermal vapour ablation therapy in the management of heterogeneous emphysema. Eur Respir J. 2012 Jun;39(6):1326-33. doi: 10.1183/09031936.00092411. Epub 2011 Nov 10. PMID 22075481